CLINICAL TRIAL: NCT06643988
Title: Neurobiological Correlates of Autobiographical Memory Training to Improve Opioid Use Disorder Outcomes
Brief Title: Autobiographical Memory in Opioid Use Disorder
Acronym: NAMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 856848
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (No Intervention): Participants who meet criteria as healthy volunteers, will receive no MemFlex training but will undergo assessments as well as fNIRS computerized tasks.
- OUD (Experimental): Participants who meet criteria for OUD and are on a stable dose of medication assisted therapy for OUD will be trained in memory flexibility training (MemFlex) - cognitive training exercises.
  Interventions: Behavioral: MemFlex

INTERVENTIONS:
Behavioral: MemFlex — MemFlex employs cognitive training exercises in self-led sessions to improve 1) switching between specific and general AMs, 2) access to positive AMs, and 3) vividness of positive AMs.
  Arms: OUD

SUMMARY:
The research study is being conducted to better understand memory function in people with opioid use disorder (OUD) and whether memory training can improve the symptoms and lives of people with OUD. Further, this study seeks to identify how brain and heart activity contribute to memory function and OUD symptoms. Participants will be asked to complete a baseline assessment, four weeks of at-home memory training (MemFlex), and a post-treatment follow-up assessment. Everyone enrolled will receive MemFlex as there is no placebo group. Each visit will include collection of a urine sample for drug testing. During the baseline and follow-up assessments, researchers will collect brain information using functional near-infrared spectroscopy (fNIRS) and heartbeat data using a wearable wristband sensor. MemFlex is a cognitive-behavioral intervention that does not pose any risk. However, the use of MemFlex in this study is experimental as it has not been tested in individuals with OUD. We will enroll 20 participants with OUD and 10 participants meeting healthy volunteer criteria.

DETAILED DESCRIPTION:
In this study, we propose to characterize possible OUD-related dysfunction in AM. We will further examine the impact of a cognitive training intervention (Memory Flexibility Training [MemFlex]) on AM and drug use outcomes and explore the underlying brain and physiological mechanisms.

Autobiographical memory and OUD:

AMs are episodic memories of one's own life. Under healthy circumstances, AMs are not simple facts (frozen in time) but are influenced by the current context to help maintain a positive sense-of-self and motivate adaptive behaviors. That is, individuals flexibly focus AM to retrieve details that help with current goals, or they adjust AM-related emotions to assist in current regulation of emotion. Patients across psychiatric disorders often have difficulty recalling specific AMs (i.e., those of a single brief event) and show dysfunction in the vividness and emotionality of AMs. The few studies on AM in OUD indicate these individuals recall fewer specific AMs have easier access to neutral AMs, and less positive AMs.

Memory Flexibility Training:

MemFlex employs cognitive training exercises in self-led sessions to improve 1) switching between specific and general AMs, 2) access to positive AMs, and 3) vividness of positive AMs. In trials for depression and posttraumatic stress, MemFlex has improved symptoms and AM recall but MemFlex has not been tested for OUD. Previous research has shown that chronic drug use can lead to increased dopaminergic brain response to drug reward cues/reminders (which are learned over time) and reduced dopaminergic brain response to receiving both drug and non-drug rewards (in-the-moment). This can create reward inflexibility, in which drug rewards drive motivation while non-drug rewards contribute relatively little. Further, work in our lab and others has shown OUD is associated with cognitive inflexibility, which is an impaired ability to switch between mental tasks when contexts change and may impair decision-making. Inflexibility in the reward and cognitive systems may leave individuals 'stuck' choosing drug rewards to the exclusion of other rewards (e.g., relationships, work). We propose that MemFlex, by improving access to non-drug reward-related AMs and the ability to switch between types of AMs, will help patients with OUD use AM to regulate emotions and pursue healthier rewards.

Neurobiological Foundation of Flexibility:

The brain's prefrontal cortex (PFC) is critical to successful cognitive flexibility and reward function. It is also implicated in AM deficits and is impaired in people with OUD. As such, we will use PFC activity during AM and reward flexibility task may explain the neural foundations of related deficits. Previous research has also shown that physiological arousal, as measured by heart rate variability (HRV), contributes to cognitive flexibility and correlates with PFC and subcortical brain areas that support flexibility. Therefore, HRV (i.e., the time fluctuation between heartbeats) may contribute to deficits in AM and reward flexibility and be a marker of MemFlex treatment success.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 60 years old.
2. Willingness to provide signed, informed consent and commit to completing study procedures
3. Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures, and must have access to a cellphone.
4. OUD subjects: Lifetime self-reported history of OUD (according to DSM-5 criteria)
5. OUD subjects: On a stable dose (at least 2 weeks without change) of MOUD (e.g., buprenorphine, methadone) as confirmed by self-report, urine drug screening, and/or the Prescription Drug Monitoring Program database.
6. OUD subjects: Access to a stable residence or space to complete the at-home treatment module

Exclusion Criteria:

1. Current severe psychiatric (e.g., bipolar disorder) or physical (e.g., dementia, Parkinson's disease) determined by self-reported history or physical exam and disorder deemed by PI to significantly interfere with brain function or make the study hazardous for the subject.
2. Head trauma or injury deemed by PI as likely to impact the prefrontal cortex (e.g., loss of consciousness for more than 30 minutes or skull fracture, intracranial bleeding, or abnormal MRI) as determined by self-reported history or physical exam.
3. Medical condition or medical treatment that may interfere with the subject's ability to complete the intervention, at discretion of the PI (e.g., extended surgery planned or expecting to give birth during the course of the study)
4. Inability to sit upright while remaining relatively still and operating a mouse and keypad.
5. Current ongoing participation in a research study or participation in a clinical trial and receipt of investigational drug(s) or intervention during 30 days prior to the research study, except as explicitly approved by the Principal Investigator.
6. Currently prescribed opioid medication for treatment of pain or other disorder (besides opioid use disorder).
7. OUD subjects: Past 1-year history of non-OUD substance use disorder (other than nicotine, alcohol, or cannabis use disorders).
8. OUD subjects: Positive urine drug screen for any tested substances except for opioids, cocaine, and cannabis at screening or the baseline assessment visit (a test may be repeated if it is needed to confirm accuracy).
9. HC subjects: Lifetime history of any substance use disorder (other than nicotine use disorder at any time and alcohol or cannabis use disorders more than 1 year ago).
10. HC subjects: Positive urine drug screen for any tested substances at screening or the baseline assessment visit (a test may be repeated if it is needed to confirm accuracy).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Autobiographical Memory (AM) Recall (AMT-AI) | Pre and Post treatment assessment (weeks 1 and 5)
  Specificity [specific vs. general] and valence [positive, negative, neutral] and PFC activity during AM recall.The AMT-AI outcomes will be the proportion of specific AMs in each condition (neutral, positive, negative) and mean ΔHbO in the mPFC and dlPFC (separately) during AM recall relative to the control block.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No